CLINICAL TRIAL: NCT05352737
Title: A Retrospective Study Exploring the Role of Serum Methylmalonic Acid (MMA) in Breast Cancer---focusing on Metastasis, Chemotherapy Resistance, and Ageing Effects
Brief Title: Exploring the Role of Serum Methylmalonic Acid (MMA) in Breast Cancer
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Qi Wu, Dr., KU Leuven
Other Study IDs: S64752
Record Dates: First submitted 2022-04-22; First posted 2022-04-29 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — peripheral serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Pri-Meta: patients with breast cancer metastasis at first diagnosis
  Interventions: Diagnostic Test: methylmalonic acid testing
- Sec-Meta: patients with early breast cancer developed distant metastasis within 5 years
  Interventions: Diagnostic Test: methylmalonic acid testing
- Non-Meta: patients with early breast cancer did not develop distant metastasis within 5 years
  Interventions: Diagnostic Test: methylmalonic acid testing
- older: patients with breast cancer older than 70 years old with G8 screening
  Interventions: Diagnostic Test: methylmalonic acid testing
- pCR: patients with breast cancer reached pCR after neoadjuvant chemotherapy
  Interventions: Diagnostic Test: methylmalonic acid testing
- non-pCR: patients with breast cancer did not reach pCR after neoadjuvant chemotherapy
  Interventions: Diagnostic Test: methylmalonic acid testing

INTERVENTIONS:
Diagnostic Test: methylmalonic acid testing

SUMMARY:
This project aims to investigate the role of MMA in breast cancer. To this end, we will measure MMA on serum samples collected at the time of breast cancer diagnosis, to investigate the role of MMA in predicting long-term recurrence risk, response to neoadjuvant chemotherapy, and its association with age and clinical frailty.

DETAILED DESCRIPTION:
This project aims to investigate the role of MMA in breast cancer. To this end, we will measure MMA on serum samples collected at the time of breast cancer diagnosis, to investigate the role of MMA in predicting long-term recurrence risk, response to neoadjuvant chemotherapy, and its association with age and clinical frailty. If the role of baseline serum MMA in therapy resistance and/or metastasis is confirmed, our study could be further extended by evaluating SOX4 expression in the tumor tissues (SOX4 is activated by MMA, and SOX4 induces EMT (epithelial to mesenchymal transition) and the metastasis process.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients older than 18 years at diagnosis.
2. First diagnosis of invasive breast cancer.
3. All pathological parameters are available to identify histological subtype according to standard procedures.
4. Availability of frozen serum samples at diagnosis.
5. Voluntarily signed Informed Consent obtained before blood drawing for biobanking was performed.

Exclusion Criteria:

1. Pregnant at diagnosis.
2. stage 0 disease (in situ).
3. Bilateral BC at diagnosis or multifocal unilateral BC with different histology.
4. Other subtypes than Invasive ductal carcinoma.
5. Prior breast cancer.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: patients with breast cancer admitted into University of Hospital, Leuven, from 2003 to 2015.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
MMA levels | baseline
  baseline serum MMA levels in pre-defined patients

CONTACTS AND LOCATIONS:
Overall Officials: Hans Wildiers, PhD, Principal Investigator — UZ Leuven
Locations (1):
- Lab of Experimental Oncology, Leuven, State Or Province:, Belgium

IPD SHARING:
Plan to Share IPD: No